CLINICAL TRIAL: NCT00843765
Title: Program of TCM on Early Rehabilitation and Secondary Prevention of Ischemic Stroke
Brief Title: Efficiency Study of Traditional Chinese Medicine (TCM) Versus Western Medicine (WM) on Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007AA02Z4B2
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Stroke
Keywords: Stroke; Traditional Chinese Medicine; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy; Massage; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM integrated group (Active Comparator): 800 patients with acupuncture, massage and basic Chinese medicine treatment
  Interventions: Other: acupuncture, massage and basic TCM treatment
- Western Medicine group (Active Comparator): 400 patients with modern rehabilitation techniques and Western Medicine basic treatment
  Interventions: Other: rehabilitation and WM basic treatment

INTERVENTIONS:
Other: acupuncture, massage and basic TCM treatment — 1. During hospitalization:Patients accept TCM rehabilitation and basic treatment including WM basic treatment and Chinese medicine injection,decoction,herb soak treatment and health education.
  2. After discharge from hospital: In the TCM group,add prescriptions according to two conditions:a. patients using A injection (one Chinese herb injection admitted by SFDA) will take A' capsule (one Chinese herb capsule admitted by SFDA) for 6 months;b.patients using B injection (ditto) will take B' capsule (ditto) for 6 months.Both of them will accept TCM health education.In the WM group, patients are suggested with targeted rehabilitation programs according to different causes.
  Other Names: 863 TCM project for ischemic stroke-TCM group
  Arms: TCM integrated group
Other: rehabilitation and WM basic treatment — there two steps:
  1. during hospitalization: patients accept modern rehabilitation and basic treatment of life supporting and medicine using and health education
  2. After discharge: make rehabilitation plans for patients including management of anticoagulant drugs, blood pressure, blood lipid and blood glucose, health education, and some suggestions for resisting alcohol ,smoking and reasonable diet
  Other Names: 863 TCM project for ischemic stroke-WM group
  Arms: Western Medicine group

SUMMARY:
Complex project of Traditional Chinese Medicine (TCM) with Western Medicine (WM) project under stroke unit mode contrast,assuming that the efficiency of TCM on early rehabilitation and secondary prevention of ischemic stroke is same or better than that of WM.

DETAILED DESCRIPTION:
As a multi-site randomized controlled clinical trial,through a central system,patients were randomly assigned to the intervention group or the control group.In the intervention group, patients were treated with the traditional Chinese medicine comprehensive rehabilitation program, which includes traditional Chinese medicine syndrome differentiation herbs, Chinese medicine injection, wash foam Chinese medicine, acupuncture,massage, and Chinese medicine health education. In the control group, patients were treated with Western-based treatment plus modern rehabilitation techniques.All patients were treated for 2 weeks. At the first day after the treatment and the 14 days after treatment, each patient was evaluated for the following three clinical indications: (1)evaluation of neurological deficits by U.S. National Institutes of Health Stroke Scale (NIHSS);(2) evaluation of motor function by the short form Fugl-Meyer motor function scoring system (FMI); and (3) assessment of limb spasticity by the modified Ashworth spasticity rating scale.

ELIGIBILITY:
Inclusion Criteria:

* According with the stroke diagnosis of Traditional Chinese Medicine
* According to atherosclerotic thrombotic cerebral infarction from Western diagnosis such as medical history and CT / MRI examinations
* It has attacked in 7 days
* The assessment of scale of NIHSS:4-24 points
* Age: ≥ 35 years and ≤ 75 years
* Patients or their legal guardians sign informed consent form

Exclusion Criteria:

* The patients with ICH or cerebral hemorrhage or TIA
* It has attacked beyond 7 days
* Patients with stroke history and the mRS ≥ 2 points before this attack
* Mixed type of stroke (infarction after bleeding or bleeding after infarction)
* Patients with cerebral infarction by cardiogenic embolism, blood hypercoagulable state and tunica intima exfoliating
* Patients with serious heart disease;failure of heart or liver or kidney; cancer;digestive tract bleeding
* Women of pregnancy or breast-feeding
* Patients who are taking part in other clinical trials that will influence the results of this study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1151 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
NIHSS Stroke Scale, relapse rate | 360 days

SECONDARY OUTCOMES:
adverse event | 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Xie Y m, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Langhorne P, Ramachandra S; Stroke Unit Trialists' Collaboration. Organised inpatient (stroke unit) care for stroke: network meta-analysis. Cochrane Database Syst Rev. 2020 Apr 23;4(4):CD000197. doi: 10.1002/14651858.CD000197.pub4. PMID 32324916